CLINICAL TRIAL: NCT04706065
Title: Genetic Polymorphisms of Serine Hydroxylmethyl Transferase 1 (SHMT1) in Patients With Parkinson's Disease
Brief Title: SHMT1 Polymorphism in Parkinson's Disease,
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Collaborators: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Effat AETony, MD, professor of internal medicine, Assiut University
Other Study IDs: aswan
Record Dates: First submitted 2021-01-03; First posted 2021-01-12 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Study the Role of SHMT1 Polymorphism in Parkinson Disease
Keywords: SHMT1 polymorphism; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP 1: Group 1 (patients with PD) All participants will be subjected to thorough history taking, full clinical and neurological examination. Diagnosis of PD by using Brain Bank Criteria for diagnosis of Parkinson Disease , assessment of the severity of PD by using PDRS and evaluation of cognitive functions using MMSE.
  Interventions: Genetic: SHMT1 polymorphism
- Group 2: Group 2 (controls) All participants will be subjected to thorough history taking, full clinical and neurological examination.
  Interventions: Genetic: SHMT1 polymorphism

INTERVENTIONS:
Genetic: SHMT1 polymorphism — It is to identify the role of SHMT1polymorphism in PD and examine the relationship between it and Severity of PD.

SUMMARY:
Parkinson Disease (PD) is the most common movement disorder and represents the second most common degenerative disease of the central nervous system . SHMT has been shown to be associated with various diseases.

DETAILED DESCRIPTION:
This case -control observational prospective study will conducted on 40 patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 50 years.
* Patients with PD diagnosed according to the United Kingdom Parkinson's Disease Society Brain Bank (UK PDS Brain Bank diagnostic criteria)

Exclusion Criteria:

* Patients with parkinsonian plus syndrome

  * Patients with secondary parkinsonism
  * Patients with other chronic comorbidities (renal, hepatic, and endocrinal disturbances and chronic chest disease.)
  * Past and /or present history of epilepsy.
  * Patients with disturbed conscious level.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient with parkinson diisease
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
polymorphism of SHMT1gene | one year

SECONDARY OUTCOMES:
the role of SHMT1plymorphism in pathogenesis PD | one year
Study the relationship of Shmt1 polymorphism to the severity of Parkinson disease | One year

CONTACTS AND LOCATIONS:
Overall Officials: Abeer a tony, MD, Principal Investigator — Assistant professor
Locations (1):
- Effat abdelhady tony, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided